CLINICAL TRIAL: NCT00204009
Title: Population-based Epidemiologic Study of Childhood Diabetes in Chicago: a) Disease Surveillance; b) Family Studies; c) Questionnaire Followup.
Brief Title: Chicago Childhood Diabetes Registry
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: R01DK044752 (NIH); IRB Protocol #s:; 11348B;; 11564B;; 12323B
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus
Keywords: children and adolescents; epidemiology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only

INTERVENTIONS:
Behavioral: Disease Surveillance, Family Studies, Questionnaire Followup

SUMMARY:
The goal of this study is to investigate the epidemiology and natural history of childhood-onset diabetes, whether of autoimmune, non-autoimmune, or mixed etiology in affected probands and their relatives.

DETAILED DESCRIPTION:
The goal of this study is to investigate the epidemiology and natural history of childhood-onset diabetes, whether of autoimmune, non-autoimmune, or mixed etiology in affected probands and their relatives. The following hypotheses frame the research questions to be addressed:

Hypothesis 1. Diabetes as it occurs in youth derives from a spectrum of etiologic processes, from the insulinopenia of autoimmune type 1 to obesity-related, insulin-resistant type 2 diabetes. A subset of children develop diabetes through a combination of the 2 major etiologic pathways, with autoimmune ß-cell destruction aggravated by the presence of insulin resistance related to genetic susceptibility, obesity and/or physical inactivity. A fraction of young patients are unclassifiable at onset due to severe symptomatology and ambiguities in measures of ß-cell function. This poses the research challenge of misclassification of disease, as well as the clinical difficulty of potentially inappropriate treatment … Since patients are drawn from the city-wide registry, clustering of genetic and behavioral risk factors will be systematically identified without the selection bias inherent in case series and clinic-based studies.

Research questions:

1. Is it feasible to distinguish type 1 from early-onset type 2 diabetes at diagnosis? Which demographic, clinical, and family characteristics are most useful?
2. Is the risk of developing diabetes among siblings of early-onset type 2 or mixed cases equivalent to that for siblings of type 1 patients? Which characteristics are most predictive of risk? Hypothesis 2. Changes in the epidemiologic parameters of childhood diabetes over the past 2 decades are directly related to changes in the prevalence of risk factors for both type 1 and type 2 diabetes, including obesity, physical inactivity, and perinatal exposures.

Research questions:

1. Is change in the incidence of childhood diabetes occurring uniformly across all age-, sex- and ethnic strata?
2. Are secular changes in type 2 incidence rates continuing, and is this occurring in all age-, sex- and ethnic strata? Hypothesis 3. A complex interplay of heritable, behavioral, and treatment factors can accelerate or delay the development of chronic diabetes complications. It is particularly compelling to understand this process in young patients, those with the most years of productive life at risk. … Recent observations indicate that features of the metabolic syndrome, over and above glycemic control, are potent risk factors for macrovascular complications. Familial aggregation of these traits may itself play a role in determining the risk of chronic complications among young people with diabetes.

Research questions:

1. Do young people with diabetes who demonstrate signs and symptoms of early complications have greater insulin resistance or other characteristics that distinguish them from those patients who are free of complications, controlled for disease duration and metabolic control?
2. Do young patients with early signs/symptoms of complications have more parents who themselves have elevated cardiovascular disease risk factors, than patients who are free of chronic complications, controlled for disease duration and metabolic control?

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with diabetes before age 18 AND resident of the City of Chicago at diagnosis

Exclusion Criteria:

* diabetes secondary to another condition, e.g. cystic fibrosis

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: target all diagnosed with diabetes before age 18 AND resident of the City of Chicago at diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 1992-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Lipton, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Biological Sciences Division, Pritzker School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Result] Lipton RB, Drum M, Burnet D, Rich B, Cooper A, Baumann E, Hagopian W. Obesity at the onset of diabetes in an ethnically diverse population of children: what does it mean for epidemiologists and clinicians? Pediatrics. 2005 May;115(5):e553-60. doi: 10.1542/peds.2004-1448. PMID 15867020
- [Result] Grover V, Lipton RB, Sclove SL. Seasonality of month of birth among African American children with diabetes mellitus in the city of Chicago. J Pediatr Endocrinol Metab. 2004 Mar;17(3):289-96. doi: 10.1515/jpem.2004.17.3.289. PMID 15112905
- [Result] Lipton RB, Zierold KM, Drum ML, Klein-Gitelman M, Kohrman AF. Re-hospitalization after diagnosis of diabetes varies by gender and socioeconomic status in urban African-American and Latino young people. Pediatr Diabetes. 2002 Mar;3(1):16-22. doi: 10.1034/j.1399-5448.2002.30104.x. PMID 15016170
- [Result] Onyemere KU, Lipton RB. Parental history and early-onset type 2 diabetes in African Americans and Latinos in Chicago. J Pediatr. 2002 Dec;141(6):825-9. doi: 10.1067/mpd.2002.130261. PMID 12461500
- [Result] Lipton RB, Drum M, Li S, Choi H. Social environment and year of birth influence type 1 diabetes risk for African-American and Latino children. Diabetes Care. 1999 Jan;22(1):78-85. doi: 10.2337/diacare.22.1.78. PMID 10333907